CLINICAL TRIAL: NCT04668729
Title: Effects of Lumbosacral Chiropractic Spinal Manipulative Therapy on Muscle Strength, Range of Motion, Balance and Pain in Olympic Style Weightlifting Athletes
Brief Title: Effects of Lumbosacral Chiropractic on the Olympic Style Weightlifting Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan Altunok, Physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1801408
Record Dates: First submitted 2020-12-05; First posted 2020-12-16 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Athletic Injuries
Keywords: Athletes; Balance; Muscle strenght; Musculoskeletal manipulations; Pain; Range of motion
MeSH Terms: conditions — Athletic Injuries; Pain | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: The individuals are randomly allocated into control and chiropractic groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 20 people will be included in the control group. 3 measurements will be taken one week apart in total. Measurements will consist of maximum isometric muscle strength, lumbar range of motion, balance performance, and pain intensity. And it will be evaluated respectively by back dynamometer, hand finger-to-ground distance (HFGD) and Modified Schober test, flamingo balance test, and visual analog scale.
- Chiropractic group (Experimental): 20 people will be included in the experimental group. Lumbal chiropractic HVLA (High Velocity, Low amplitude: HVLA) spinal manipulation and sacroiliac joint chiropractic HVLA manipulation will be applied 3 times in total with a weekly interval. The maximum isometric muscle strength before and immediately after the application, lumbar joint range of motion, balance performance, and pain intensity will be evaluated respectively by back dynamometer, hand finger-to-ground distance (HFGD), and Modified Schober test, flamingo balance test, and visual analog scale.
  Interventions: Other: Chiropractic Manipulation

INTERVENTIONS:
Other: Chiropractic Manipulation — Lumbar vertebrae and sacroiliac joints of the participants that have lost their normal joint motion will be detected by static and dynamic palpation techniques.
  Lumbal Chiropractic HVLA Spinal Manipulation: HVLA manipulation will be applied in the left transverse process of the lumbar vertebra (mammillary process) of the participants whose problem is to the left of the lumbar vertebra.
  Sacroiliac Chiropractic HVLA Manipulation: Participants who lost normal joint motion in the anterior and superior directions in the left sacroiliac joint will be treated with HVLA manipulation in the left PSIS (Posterior Superior Iliac Spine: PSIS). Participants who have lost normal joint motion in the left sacroiliac joint in the posterior and inferior directions will be applied HVLA manipulation in the left ischial tuberosity.
  For both applications, it will be positioned in the opposite position for the problems on the right and the application will be made in the opposite position.
  Arms: Chiropractic group

SUMMARY:
It is known that low back injuries experienced by weightlifting athletes cause a decrease in performance. The effects of spinal manipulative therapy, which has been found to positively affect performance in various sports, are not known in the Olympic style weightlifting athletes. This study is aimed to investigate the effects of lumbosacral chiropractic spinal manipulative therapy on muscle strength, range of motion, balance, and pain in Olympic style weightlifting athletes.

In this research, 40 male Olympic style weightlifting athletes are planned to take place. Male athletes will be randomly divided into two groups as a control and a treatment group. To the individuals in the treatment group; lumbal region chiropractic high-speed, low amplitude (High Velocity, Low amplitude: HVLA) spinal manipulation and sacroiliac joint chiropractic HVLA manipulation are planned to perform once a week for a total of three weeks. No manipulation will be made to individuals in the treatment group. Before and after the manipulation; the maximum isometric muscular force, the lumbar spine range of motion, balance performance and pain intensity will be evaluated by a back dynamometer, hand finger-ground distance test (HFGD), and Modified Schober test, flamingo balance test, and visual analog scale. SPPS 25 (IBM Corp. Released 2017. IBM SPSS Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp.) version will be used to analyze the data.

DETAILED DESCRIPTION:
There are studies in the literature regarding the positive effect of chiropractic treatment on musculoskeletal injuries. In a study, it is found that the group that received cervical chiropractic manipulation on judo athletes showed a statistically significant (p <0.05) increase in grip strength compared to those who received sham practice. In another study, it is found that a single lumbar spinal manipulation reduced the relative strength difference between the limbs for knee and hip flexion (p <0.05). In another study, it is shown that a single spinal manipulation session increased the muscle strength of the ankle plantar flexor muscles and corticospinal excitability (p <0.05) in elite Taekwondo athletes. Likewise, according to another study, lumbopelvic joint manipulation increased quadriceps activation and strength.

A study claims that young female athletes with talocrural joint dysfunction showed a statistically significant (p <0.05) improvement in vertical jump height after chiropractic manipulation. In addition, in a study investigating the effect of pelvic manipulation on vertical jump height in female university students with functional leg length inequality, it was found that after the intervention, jump height improved significantly only in the pelvic manipulation group compared to pre-intervention height, while improvement in female university students with functional leg length inequality was found to be statistically significant (p <0.05) in both manipulation and stretching groups after the manipulation.

A study showed that chiropractic spinal manipulative therapy can increase hip extension ability in young running athletes (p <0.05). According to a study conducted on football players, it was shown that combined manipulative interventions caused significantly (p <0.05) increases in the range of motion in the lumbar region and sacroiliac joint flexion. In addition, it was reported that the group who received chiropractic manipulation (compared to the group that received sham manipulation) caused a significant increase in kick speed (p <0.05) after the manipulation.

Again, in another research, it is found that an increase in cervical range of motion and a decrease in neck pain with a single cervical HVLA (High Velocity, Low amplitude: HVLA) manipulation (p <0.05) and stated that HVLA manipulation was more effective than mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Being a weightlifting athlete
* Presence of sacroiliac and lumbar spine asymptomatic dysfunctions in tests

Exclusion Criteria:

* Not wanting to continue education
* Not being able to come to assessments
* Having a musculoskeletal injury in the upper and lower extremities in the last month
* Having any neurological or psychiatric illness
* Having a fracture in the past
* Having a tumor in the past
* Lumbar disc hernias, spondylosis, spondylolisthesis
* Having a disease related to the cardiac and respiratory system
* Having an infectious, rheumatological, metabolic, and endocrine disease
* Having dislocation, osteoporosis, ankylosing spondylitis, discopathy, rheumatoid arthritis
* Being in the treatment of instability, acute myelopathy, anticoagulants
* Recently had a surgery

Ages: 13 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 3 weeks
  Muscle Strength: In measuring the muscle strength of the back area, the participant will be provided to take the starting position for the test on the dynamometer (Takkei-Japon) while the knees are flexed. Then, while his/her arms are in extension, his/her back is straight, and his/her body is slightly flexed, he/she will be asked to pull up the dynamometer bar he grasped with his/her hands vertically using his legs at the maximum level. This traction will be repeated three times. The best result will be recorded.
Lumbal Area Joint Range of Motion: Hand Finger-Ground Distance (HFGD) | 3 weeks
  Hand Finger-Ground Distance (HFGD): Participants will lean forward as much as they can, standing, hands-free, without bending their knees. Lumbar joint range of motion will be found by measuring the distance between the participants' third finger and the ground.
Lumbal Area Joint Range of Motion: Modified Schober Test | 3 weeks
  Modified Schober Test: With the participants standing in an upright position, a line will be drawn joining the right and left posterior superior iliac spine. From the midpoint of this line, 10 cm up and 5 cm below will be marked, the participants will be asked to lean forward as much as possible without bending their knees, and the distance between the two will be measured again. Lumbal joint range of motion will be obtained by recording the measured value above 15 cm as a result of the modified Schober test.
Balance Performance | 3 weeks
  Flamingo balance test: Specially prepared balance bench (fifty cm long, four cm high, three cm wide) and timekeeper will be used in the test. The participant will be placed on the balance bench with his dominant foot. Then, the participant will be asked to flex the other knee, pull it towards the hip and hold it with the same hand. After the participant takes the correct position, s/he will get help from the test manager by holding on to the test manager until he/she stabilizes, and the time will start from the moment he/she stabilizes and quits the support. The time will be stopped when the participant's balance is disrupted, that is, when s/he leaves his/her foot, falls from the bench, any part of the body touches the ground, and so on. The total time will be a minute. The number of times the participants are unbalanced during the test (falling etc.) will be counted and recorded as the athletes' scores at the end of the test. Low scores mean better, higher scores mean worse outcome.
Pain Intensity | 3 weeks
  Pain Intensity: It will be evaluated with a visual analog scale (VAS) numbered equal intervals from 0 to 10 on a 10 cm line, which is used to digitize some values that cannot be measured numerically. 0 means no pain and 10 means unbearable pain. Thus, participants will be asked to mark the intensity of pain they perceive.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ataş Balcı, assist prof, Study Director — Bahçeşehir University; Kenan Erdağı, assist prof, Study Director — Necmettin Erbakan University
Locations (1):
- Ankara Türkiye Olimpiyat Hazirlik Merkezi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botelho MB, Andrade BB. Effect of cervical spine manipulative therapy on judo athletes' grip strength. J Manipulative Physiol Ther. 2012 Jan;35(1):38-44. doi: 10.1016/j.jmpt.2011.09.005. Epub 2011 Nov 10. PMID 22079053
- [Background] Chilibeck PD, Cornish SM, Schulte A, Jantz N, Magnus CR, Schwanbeck S, Juurlink BH. The effect of spinal manipulation on imbalances in leg strength. J Can Chiropr Assoc. 2011 Sep;55(3):183-92. PMID 21886280
- [Background] Christiansen TL, Niazi IK, Holt K, Nedergaard RW, Duehr J, Allen K, Marshall P, Turker KS, Hartvigsen J, Haavik H. The effects of a single session of spinal manipulation on strength and cortical drive in athletes. Eur J Appl Physiol. 2018 Apr;118(4):737-749. doi: 10.1007/s00421-018-3799-x. Epub 2018 Jan 11. PMID 29327170
- [Background] Grindstaff TL, Hertel J, Beazell JR, Magrum EM, Ingersoll CD. Effects of lumbopelvic joint manipulation on quadriceps activation and strength in healthy individuals. Man Ther. 2009 Aug;14(4):415-20. doi: 10.1016/j.math.2008.06.005. Epub 2008 Sep 20. PMID 18805726
- [Background] Hedlund S, Nilsson H, Lenz M, Sundberg T. Effect of chiropractic manipulation on vertical jump height in young female athletes with talocrural joint dysfunction: a single-blind randomized clinical pilot trial. J Manipulative Physiol Ther. 2014 Feb;37(2):116-23. doi: 10.1016/j.jmpt.2013.11.004. Epub 2014 Jan 2. PMID 24387886
- [Background] Gong W. The influence of pelvic adjustment on vertical jump height in female university students with functional leg length inequality. J Phys Ther Sci. 2015 Jan;27(1):251-3. doi: 10.1589/jpts.27.251. Epub 2015 Jan 9. PMID 25642085
- [Background] Sandell J, Palmgren PJ, Bjorndahl L. Effect of chiropractic treatment on hip extension ability and running velocity among young male running athletes. J Chiropr Med. 2008 Jun;7(2):39-47. doi: 10.1016/j.jcme.2008.02.003. PMID 19674719
- [Background] Deutschmann KC, Jones AD, Korporaal CM. A non-randomised experimental feasibility study into the immediate effect of three different spinal manipulative protocols on kicking speed performance in soccer players. Chiropr Man Therap. 2015 Jan 13;23(1):1. doi: 10.1186/s12998-014-0046-3. eCollection 2015. PMID 25635222
- [Background] Martinez-Segura R, Fernandez-de-las-Penas C, Ruiz-Saez M, Lopez-Jimenez C, Rodriguez-Blanco C. Immediate effects on neck pain and active range of motion after a single cervical high-velocity low-amplitude manipulation in subjects presenting with mechanical neck pain: a randomized controlled trial. J Manipulative Physiol Ther. 2006 Sep;29(7):511-7. doi: 10.1016/j.jmpt.2006.06.022. PMID 16949939